CLINICAL TRIAL: NCT05542004
Title: Nationwide Utilization of Danish Government Electronic Letter System for Increasing InFLUenza Vaccine Uptake
Acronym: NUDGE-FLU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tor Biering-Sørensen (Other)
Collaborators: Statens Serum Institut (Other); Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor-Investigator, Tor Biering-Sørensen, Professor, MD, PhD, MPH, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FLU00180
Record Dates: First submitted 2021-08-31; First posted 2022-09-15 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Influenza; Behavior and Behavior Mechanisms
Keywords: Influenza; Vaccination; Nudging; Behavioral Science
MeSH Terms: conditions — Influenza, Human; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Control (No Intervention): No letter
- Standard Letter (Experimental): This group will receive a standard letter on the benefits of influenza vaccination without behavioral economic enhancement
  Interventions: Behavioral: Behavioral Economic Principles
- Priming & Hot State Activation - 1 reminder (Experimental): The standard letter sent out two times instead of once
  Interventions: Behavioral: Behavioral Economic Principles
- Depersonalized Letter (Experimental): The standard letter without the recipient's name
  Interventions: Behavioral: Behavioral Economic Principles
- Gain-Framing/Context (Experimental): Text added to the standard letter employing the specified behavioral economic principle
  Interventions: Behavioral: Behavioral Economic Principles
- Loss-Framing/Context (Experimental): Text added to the standard letter employing the specified behavioral economic principle
  Interventions: Behavioral: Behavioral Economic Principles
- Collective Goal (Experimental): Text added to the standard letter employing the specified behavioral economic principle
  Interventions: Behavioral: Behavioral Economic Principles
- Active Choice/Implementation Intention Prompt (Experimental): Text added to the standard letter employing the specified behavioral economic principle
  Interventions: Behavioral: Behavioral Economic Principles
- Cardiovascular Gain Frame (Experimental): Text added to the standard letter employing the specified behavioral economic principle
  Interventions: Behavioral: Behavioral Economic Principles
- Expert Authority (Experimental): Text added to the standard letter employing the specified behavioral economic principle
  Interventions: Behavioral: Behavioral Economic Principles

INTERVENTIONS:
Behavioral: Behavioral Economic Principles — The control arm will receive no letter to reflect the background vaccination uptake. Intervention arms will test the effects of different letters developed using behavioral economic principles.
  Arms: Active Choice/Implementation Intention Prompt; Cardiovascular Gain Frame; Collective Goal; Depersonalized Letter; Expert Authority; Gain-Framing/Context; Loss-Framing/Context; Priming & Hot State Activation - 1 reminder; Standard Letter

SUMMARY:
In randomized clinical trials and observational studies, influenza vaccination has been shown to be effective in reducing influenza-related illness, hospitalizations, cardiovascular events, and mortality in select populations. However, the real-world effectiveness of influenza vaccination is limited by its uptake. This study will investigate investigate whether digital behavioral nudges delivered via the official, mandatory Danish electronic letter system can increase influenza vaccine uptake among eligible influenza vaccination candidates.

DETAILED DESCRIPTION:
The study is a prospective, randomized, open-label implementation trial. The study population will consist of persons identified as eligible for free-of-charge influenza vaccination in the Danish health system aged 18 years and above. Subjects will be identified through Danish nationwide health registries using codes from the International Classification of Diseases, 10th revision (ICD-10) and the Anatomical Therapeutic Chemical (ATC) classification system. Individuals will be randomized to 1 of 10 arms (1 control arm and 9 intervention arms) with each testing different nudging strategies employing various behavioural economic principles. The interventions will be delivered through the official, mandatory Danish electronic letter system. All subject data will be retrieved from the Danish nationwide registries with the exception of information on intervention allocation. Endpoints will be retrieved at prespecified dates using prespecified search algorithms. The study will be performed in collaboration with the Danish Health Data Authority and Statens Serum Institut.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=65 years at January 15, 2023 (eligible for free influenza vaccination in the official Danish vaccination program)
2. Access to the official, mandatory Danish electronic mailbox system

Exclusion Criteria:

1) Persons living in nursing homes

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 964870 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Number of participants who received an influenza vaccine | Up to 3 months

SECONDARY OUTCOMES:
Time from intervention delivery to influenza vaccination | Up to 3 months

OTHER OUTCOMES:
Number of participants with laboratory-confirmed influenza | Up to 8 months
Number of participants with a hospitalization with influenza or pneumonia | Up to 8 months
Number of participants with any hospitalization | Up to 8 months
All-cause mortality | Up to 8 months
Composite of incident heart failure, heart failure hospitalization, or cardiovascular death | Up to 8 months
Composite of myocardial infarction, stroke, or cardiovascular death | Up to 8 months
Composite of myocardial infarction, coronary revascularization, stroke, or cardiovascular death | Up to 8 months
Number of participants with incident heart failure or heart failure hospitalization | Up to 8 months
Cardiovascular death | Up to 8 months
Number of participants with myocardial infarction | Up to 8 months
Number of participants with coronary revascularization | Up to 8 months
Number of participants with stroke | Up to 8 months
Number of contacts to general practitioner (excluding vaccination visit) | Up to 8 months
Number of participants with laboratory-confirmed COVID-19 | Up to 8 months
Number of participants with a hospitalization due to COVID-19 | Up to 8 months
Number of participants who received a COVID-19 vaccine | Up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Tor Biering-Sørensen, MD, PhD, MPH, Principal Investigator — Research Director
Locations (1):
- Center for Translational Cardiology and Pragmatic Randomized Trials, Department of Cardiology, Copenhagen University Hospital - Herlev and Gentofte, Hellerup, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected from Danish administrative health registries, which are subject to Danish legislation and can only be made available to a third party under certain conditions. Please contact the sponsor-investigator in case of any inquiries.

REFERENCES:
- [Derived] Bhatt AS, Johansen ND, Vaduganathan M, Modin D, Pareek M, Chatur S, Claggett BL, Janstrup KH, Larsen CS, Larsen L, Wiese L, Dalager-Pedersen M, Dueger EL, Samson S, Loiacono MM, Harris RC, Kober L, Solomon SD, Martel CJ, Sivapalan P, Jensen JUS, Biering-Sorensen T. Electronic Nudges and Influenza Vaccination Among Patients With a History of Myocardial Infarction: Insights From 3 Nationwide Randomized Clinical Trials. JAMA Cardiol. 2025 Jan 1;10(1):78-86. doi: 10.1001/jamacardio.2024.4648. PMID 39550717
- [Derived] Johansen ND, Vaduganathan M, Bhatt AS, Lee SG, Modin D, Claggett BL, Dueger EL, Samson S, Loiacono MM, Harris RC, Kober L, Solomon SD, Sivapalan P, Jensen JUS, Martel CJ, Krause TG, Biering-Sorensen T. Clinical Outcomes With Electronic Nudges to Increase Influenza Vaccination : A Prespecified Analysis of a Nationwide, Pragmatic, Registry-Based, Randomized Implementation Trial. Ann Intern Med. 2024 Apr;177(4):476-483. doi: 10.7326/M23-2638. Epub 2024 Mar 19. PMID 38498876
- [Derived] Lassen MCH, Johansen ND, Vaduganathan M, Bhatt AS, Lee SG, Modin D, Claggett BL, Dueger EL, Samson SI, Loiacono MM, Fralick M, Kober L, Solomon SD, Sivapalan P, Jensen JUS, Martel CJ, Krause TG, Biering-Sorensen T. Electronically Delivered Nudges to Increase Influenza Vaccination Uptake in Older Adults With Diabetes: A Secondary Analysis of the NUDGE-FLU Trial. JAMA Netw Open. 2023 Dec 1;6(12):e2347630. doi: 10.1001/jamanetworkopen.2023.47630. PMID 38117499
- [Derived] Johansen ND, Vaduganathan M, Bhatt AS, Lee SG, Modin D, Claggett BL, Dueger EL, Samson S, Loiacono MM, Harris RC, Kober L, Solomon SD, Sivapalan P, Jensen JUS, Martel CJ, Valentiner-Branth P, Krause TG, Biering-Sorensen T. Electronic nudges to increase influenza vaccination uptake among patients with heart failure: A pre-specified analysis of the NUDGE-FLU trial. Eur J Heart Fail. 2023 Aug;25(8):1450-1458. doi: 10.1002/ejhf.2913. Epub 2023 Jun 4. PMID 37211967
- [Derived] Johansen ND, Vaduganathan M, Bhatt AS, Lee SG, Modin D, Claggett BL, Dueger EL, Samson SI, Loiacono MM, Kober L, Solomon SD, Sivapalan P, Jensen JUS, Martel CJ, Valentiner-Branth P, Krause TG, Biering-Sorensen T. Electronic nudges to increase influenza vaccination uptake in Denmark: a nationwide, pragmatic, registry-based, randomised implementation trial. Lancet. 2023 Apr 1;401(10382):1103-1114. doi: 10.1016/S0140-6736(23)00349-5. Epub 2023 Mar 5. PMID 36889332
- [Derived] Modin D, Johansen ND, Vaduganathan M, Bhatt AS, Lee SG, Claggett BL, Dueger EL, Samson SI, Loiacono MM, Kober L, Solomon SD, Sivapalan P, Jensen JUS, Jean-Marie Martel C, Valentiner-Branth P, Krause TG, Biering-Sorensen T. Effect of Electronic Nudges on Influenza Vaccination Rate in Older Adults With Cardiovascular Disease: Prespecified Analysis of the NUDGE-FLU Trial. Circulation. 2023 May 2;147(18):1345-1354. doi: 10.1161/CIRCULATIONAHA.123.064270. Epub 2023 Mar 5. PMID 36871213
- [Derived] Johansen ND, Vaduganathan M, Bhatt AS, Lee SG, Modin D, Claggett BL, Dueger EL, Samson S, Loiacono MM, Kober L, Solomon SD, Sivapalan P, Jensen JUS, Valentiner-Branth P, Krause TG, Biering-Sorensen T. Nationwide Utilization of Danish Government Electronic letter system for increasing inFLUenza vaccine uptake (NUDGE-FLU): Study protocol for a nationwide randomized implementation trial. Am Heart J. 2023 Jun;260:58-71. doi: 10.1016/j.ahj.2023.02.009. Epub 2023 Feb 17. PMID 36801265